CLINICAL TRIAL: NCT00583895
Title: Phase IIa, Randomized, Double-blind, Placebo-controlled, Intra-individual Left-right Limb Comparison Trial in 25 Patients With Moderate Atopic Dermatitis to Investigate the Efficacy, Local Irritation, Safety, Tolerability and Pharmacokinetics of Twice Daily Topical Applications With 10% ImCOOH Cream for 14 Days With an Additional Morning Application on Day 15.
Brief Title: Safety and Efficacy Study of ImCOOH Cream in Patients Suffering From Moderate Atopic Dermatitis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recruitment problems; insufficient number of new recruits
Sponsor: Valletta Health B.V. (Industry)
Responsible Party: F. W.G. Trouwen, M.Sc., Valletta Health B.V.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VAL-UOP-C201
Record Dates: First submitted 2007-12-20; First posted 2008-01-02 (Estimated); Last update posted 2010-03-01 (Estimated); Status verified 2010-02

CONDITIONS: Atopic Dermatitis
Keywords: dermatitis; atopic; ImCOOH; safety; tolerability; efficacy; pharmacokinetics
MeSH Terms: conditions — Dermatitis, Atopic; Dermatitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Twenty patients will receive a hydrophilic cream containing 10% ImCOOH and a placebo cream randomized over both limbs twice daily for 14 days with an additional morning application on Day 15.
  Interventions: Drug: 10% ImCOOH cream
- 2 (Placebo Comparator): Five patients will receive placebo cream on both limbs twice daily for 14 days with an additional morning application on Day 15.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 10% ImCOOH cream — Twenty patients will receive a hydrophilic cream containing 10% ImCOOH and a placebo cream randomized over both limbs twice daily for 14 days with an additional morning application on Day 15.
  Arms: 1
Drug: Placebo — Five patients will receive placebo cream on both limbs twice daily for 14 days with an additional morning application on Day 15.
  Arms: 2

SUMMARY:
Atopic dermatitis is one of the most common skin diseases, with a lifetime prevalence of up to 20%, and an increasing number of cases. Although there are a variety of treatments the number of specific medications for treating this chronic disease is limited and often not helpful, especially in more severe cases. In addition,most treatments may be used only for a limited period or are less effective in the long term (tachyphylaxis). The development of new compounds is mandatory for treatment of this often chronically recurring disease. The current trial will determine the efficacy, safety and tolerability of the endogenous compound imidazole-4-carboxylic acid (ImCOOH) administered as a topical cream twice daily for 14 days in patients with atopic dermatitis.

DETAILED DESCRIPTION:
This is a Phase IIa, randomized, double-blind, placebo-controlled, intra-individual left-right limb comparison trial to investigate the efficacy, local irritation, safety, tolerability and pharmacokinetics of multiple topical applications of ImCOOH cream. The trial population will consist of 25 patients with moderate atopic dermatitis. Twenty patients will receive a hydrophilic cream containing 10% ImCOOH and a placebo cream randomized over both limbs twice daily for 14 days with an additional morning application on Day 15. Five patients will receive placebo cream on both limbs twice daily for 14 days with an additional morning application on Day 15. The creams will be applied on 2 comparative target areas (minimum 0.1% and maximum 2% of the total body surface area per target area), with one site at the left limb and one site at the right limb. The applied creams needs to be prevented from wiping off. Efficacy will be assessed until Day 15 and safety and tolerability will be monitored until 14 days after the last application.

Efficacy will be assessed by determining the Topical Atopic Dermatitis Severity Index (toADSI) score, and the Visual Analogue Scale for Pruritis (VAS) score for both target areas at screening, predose on Day 1 of treatment and on Days 2, 7, 9, 12 and 15 of treatment. In addition, color pictures of the target areas will be taken predose on Day 1 of treatment and on Days 7 and 15 of treatment. Finally the Eczema Area and Severity Index (EASI) score will be determined for both target areas, predose on Day 1 of treatment and on Days 7 and 15 of treatment.

Safety will be assessed by monitoring (S)AEs, performing clinical laboratory tests (hematology, biochemistry, urinalysis) and physical exams and by taking vital signs and recording ECGs on a regular basis.

For pharmacokinetic analysis, plasma concentrations of ImCOOH will be determined on Days 1 and 15 up to 12 hours postdose. In addition, the morning predose plasma concentration of ImCOOH will be determined on Days 2, 4, 7, 9, and 12. Full urinary output will be collected on Day 15 up to 12 hours postdose to determine the amount of unchanged ImCOOH excreted in urine. In the patients who received the placebo cream only, the endogenous ImCOOH concentrations in plasma and urine will be measured.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged between 18 and 70 years, extremes included.
2. Skin type I, II, III, or IV.
3. Able to comply with protocol requirements.
4. Informed Consent Form (ICF) signed voluntarily before the first trial-related activity.
5. Nonsmoking or smoking no more than 10 cigarettes, or 2 cigars, or 2 pipes per day for at least 3 months prior to selection.
6. Normal weight as defined by a Quetelet Index (Body Mass Index [BMI]: weight in kg divided by the square of height in meters) of 18.0 to 30.0 kg/m2, extremes included.
7. Patients having atopic dermatitis according to the integrated list with criteria for atopic dermatitis.
8. Comparative target areas: minimum 0.1% and maximum 2% of the total body surface area per target area with one site at the left limb and one site at the right limb. Both target areas should be located at the arms (armpits [axillas] are also allowed) or both target areas should be located at the hollows of the knee.
9. Topical Atopic Dermatitis Severity Index (toADSI) score of at least 5 for both target areas and the severity of the 2 sites do not differ by more than 3 points.
10. General medical condition, in the investigator's opinion, does not interfere with the assessments and the completion of the trial.

Exclusion Criteria:

1. Female subject of childbearing potential without use of effective birth control methods, or not willing to continue practicing these birth control methods for at least 30 days after the end of the treatment period;

   Note: Estrogen based hormonal contraception may not be reliable when ImCOOH cream is applied, therefore to be eligible for this trial, women of childbearing potential should either:
   1. use a double barrier method to prevent pregnancy (i.e., using a condom with either diaphragm or cervical cap);
   2. use hormonal based contraceptives in combination with a barrier contraceptive (i.e., male condom, diaphragm or cervical cap, or female condom);
   3. use an intrauterine device in combination with a barrier contraceptive (i.e., male condom, diaphragm or cervical cap, or female condom);
   4. be only non-heterosexually active, practice heterosexual abstinence, or have a vasectomized partner (confirmed sterile).

   Women with tubal ligation are required to use 1 non-hormonal contraceptive method.

   Women who are postmenopausal for at least 2 years, and women with total hysterectomy are considered of non-childbearing potential.
2. A positive pregnancy test or breast feeding at screening.
3. A positive HIV-1 or -2 test at trial screening.
4. Hepatitis B infection (confirmed by hepatitis B surface antigen) or hepatitis C infection (confirmed by hepatitis C virus antibody) at trial screening.
5. Having a target area that is hairy in such extent that in the investigator's opinion it could influence the application.
6. Having a target area that is tattooed.
7. Unable to take venous blood samples for pharmacokinetics (PK) outside the elbow fold (fossa cubitus) area in case both elbow folds are part of the target areas.
8. Patients receiving radiation therapy, systemic therapy with cytostatics or immunosuppressive drugs within 24 weeks before the first application of trial medication.
9. Patients receiving phototherapy or systemic therapy for atopic dermatitis within 4 weeks before the first application of trial medication.
10. Patients receiving antibiotics or topical therapy for atopic dermatitis within 2 weeks before the first application of trial medication. However, once-daily use of 1% hydrocortisone acetate is allowed on all lesions with the exception of the test sites and emollients are allowed to be used liberally but not on the test sites.
11. Patients taking antihistamines within 1 week before the first application of trial medication.
12. Patients with any acute skin infection (superinfection or secondary impetiginisation).
13. Any condition (including but not limited to alcohol and drug use), which in the opinion of the investigator could compromise the patient safety or compliance with trial procedures.
14. Any history or currently active allergy such as but not limited to drug allergy, food allergy or hay fever.
15. Previously demonstrated clinically significant allergy or hypersensitivity to any of the excipients of the trial medication administered in this trial.
16. Participation in an investigational drug trial within 30 days prior to the first application of trial medication.
17. Donation of blood or plasma in the 60 days preceding the first application of trial medication.
18. Patients with the following laboratory abnormalities at screening:

    * serum creatinine > 1.1 x ULN;
    * hemoglobin ≤ 10.9 g/dL;
    * platelet count grade ≤ 125 x 109/L;
    * absolute neutrophil count ≤ 1.3 x 109/L;
    * aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≥ 1.25 x ULN;
    * total bilirubin ≥ 1.1 x ULN;
    * proteinuria or hematuria;
    * any other moderate or severe laboratory abnormality.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2007-12; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Topical Atopic Dermatitis Severity Index (toADSI) score | screening, predose on Day 1 and on Day 2, 7, 9 and 15
Visual Analogue Scale for Pruritis (VAS) score | Screening, Day 1 predose, Day 2, 7, 9, 12 and 15

SECONDARY OUTCOMES:
Eczema Area and Severity Index (EASI) score | Day 1 predose, Day 7 and 15
ImCOOH plasma and urine concentrations | Day 1 and 15 (plasma) up to 12 hours postdose and predose on Day 2, 4, 7, 9 and 12. Day 15(urine) up to 12 hours postdose

CONTACTS AND LOCATIONS:
Overall Officials: Jan D Bos, M.D., Ph.D, FRCP, Study Chair — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- InPEC B.V. (Clinical Research Unit), Torremolinos, Malaga, Spain